CLINICAL TRIAL: NCT00955500
Title: Effect of the Proteins of the Diet in Patients With Cirrhosis and a Prior Episode of Hepatic Encephalopathy. A Randomized Study
Brief Title: Effects of Proteins in Patients With Cirrhosis and Prior Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Juan Córdoba, MD, Hospital Universitari Vall d´Hebron
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PR(HG)61/2002
Record Dates: First submitted 2009-07-21; First posted 2009-08-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Cirrhosis; Proteins of the diet; Branched-chain amino acids
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Amino Acids, Branched-Chain; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal-protein diet (Active Comparator): Daily diet containing 35 kcal/kg/day, 0.7 grams of proteins/kg/day + 30 grams of oral branched-chain amino acids (leucine: 13.5 grams, isoleucine: 9 grams, valine: 7.5 grams).
  Interventions: Dietary Supplement: Branched-chain amino acids
- Low-protein diet (Active Comparator): Daily diet containing 35 kcal/kg/day, 0.7 grams of proteins/kg/day + 30 grams of oral maltodextrine
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Branched-chain amino acids — 30 grams of oral branched-chain amino acids (leucine: 13.5 grams, isoleucine: 9 grams, valine: 7.5 grams) daily
  Arms: Normal-protein diet
Dietary Supplement: Maltodextrin — 30 grams of oral maltodextrin daily
  Arms: Low-protein diet

SUMMARY:
The purpose of this study is to compare a normal-protein diet containing branched-chain amino acids to a low-protein diet in patients with non-terminal cirrhosis (MELD < 25) who have developed an episode of hepatic encephalopathy within two months prior to inclusion.

DETAILED DESCRIPTION:
Hepatic encephalopathy is a major complication of cirrhosis associated with poor prognosis and poor quality of life. Appearance of HE occurs in the setting of precipitating factors that increase plasma ammonia. The gastrointestinal tract is the primary source of ammonia, which is produced by enterocytes from glutamine and by colonic bacterial catabolism of nitrogenous sources, such as ingested proteins. This is the rationale for proposing low-protein diet as strategy to reduce ammonia production and as standard diet in patients with cirrhosis and hepatic encephalopathy. However, low-protein diet could cause wasting muscle and predispose to recurrence of hepatic encephalopathy, since muscle is an important site for extrahepatic ammonia removal.

Branched-chain amino acids have shown beneficial effects on mental state of patients with chronic hepatic encephalopathy. The possible mechanism of action may be improvement of nutritional status through induction of protein synthesis. However, role of branched-chain amino acids in treatment and prevention of acute hepatic encephalopathy is not established.

Administration of a normal-protein diet containing oral branched-chain amino acids may reduce recurrence of hepatic encephalopathy as compared to a low-protein diet.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of the liver.
* Recovery from an episode of hepatic encephalopathy within two months prior to inclusion.
* Compliance with a standard diet during two weeks prior to inclusion.

Exclusion Criteria:

* End-stage cirrhosis (MELD score > 25).
* Marked cognitive disorder (mini-mental test < 27).
* Non-treatable hepatocarcinoma in accordance with Milan criteria.
* Comorbid conditions with a life expectancy less than 6 months.
* Neurological conditions that difficult assessment of treatment of hepatic encephalopathy (dementia, encephalitis, severe depression).
* Diseases requiring administration of a specific diet (malabsorption, chronic diarrhea, chronic pancreatic insufficiency, severe obesity).
* No acceptation of written consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hepatic encephalopathy-free survival | 56 weeks

SECONDARY OUTCOMES:
Overall duration in days of episodic hepatic encephalopathy | 56 weeks
Minimal hepatic encephalopathy assessed by neuropsychological tests | 56 weeks
Health-related quality of life | 56 weeks
Nutritional status | 56 weeks
Liver function | 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Córdoba, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (3):
- Spain (3):
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de Sant Pau, Barcelona